CLINICAL TRIAL: NCT01123694
Title: Xeroderma Pigmentosum: A Survey of Patient Experiences
Brief Title: Xeroderma Pigmentosum Patient Experiences
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henry Ford Health System (Other)
Responsible Party: Henry Lim, MD, Henry Ford Hospital Department of Dermatology
Other Study IDs: IRB #5672
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Xeroderma Pigmentosum
Keywords: xeroderma pigmentosum; quality of life; DLQI; CDLQI
MeSH Terms: conditions — Xeroderma Pigmentosum | interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Xeroderma Pigmentosum patients: Xeroderma Pigmentosum patients who attend Camp Sundown, a camp for children with this condition.
  Interventions: Other: Survey Study

INTERVENTIONS:
Other: Survey Study — Survey regarding quality of life

SUMMARY:
Xeroderma Pigmentosum (XP) is a rare skin condition that causes extreme sensitivity to the sun and an increased incidence of skin cancers. The purpose of this study is to find out more about XP patient experiences and their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of xeroderma pigmentosum
* Any age
* Access to a public or private computer

Exclusion Criteria:

* Patients who do not have a confirmed diagnosis of XP
* Patients under 18 who do not have a parent/guardian able to read or speak English
* Patients who are unable to read or speak English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will be a convenience sample of XP patients from Camp Sundown, a camp for children with XP.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Henry W Lim, M.D., Principal Investigator — Henry Ford Hospital Department of Dermatology
Locations (1):
- Henry Ford Medical Center, New Center One, Detroit, Michigan, United States